CLINICAL TRIAL: NCT03360201
Title: A Formative Study to Develop Culturally Valid Psychosocial Assessment Tools and Interventions to Promote Family Well-Being in Kenya - Part II
Brief Title: An Evaluation of a Family Counseling Intervention ("Tuko Pamoja") in Kenya: a Single Case Series Design
Acronym: C0058 (4A)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Moi University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0210 (4A)
Record Dates: First submitted 2017-11-01; First posted 2017-12-04 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Mental Health; Family Relations; Family Conflict; Child Mental Disorder; Adolescent - Emotional Problem; Adolescent Problem Behavior; Child Behavior; Child Abuse; Marital Conflict; Domestic Violence; Parent-Child Relations; Parenting
Keywords: Africa; Kenya; Family relations; Child mental health; Adolescent mental health; Family therapy; Program evaluation; Family Conflict; Marital Conflict; Domestic Violence; Parenting; Parent-Child Relations; child abuse; low- and middle-income country
MeSH Terms: conditions — Psychological Well-Being; Neurodevelopmental Disorders; Child Behavior

STUDY DESIGN:
Intervention Model Description: The study will follow a single case (N of 1) series design. Pre-post changes will be measured, and repeated measures will be administered before, during, and following the intervention to track change over time. The timing of entry into the study and the numbers of repeated measures data points are randomized across families. Data analysis will aim to (a) identify patterns of change over the course of the intervention and (b) relate change trajectories to theorized mechanisms of action.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: Tuko Pamoja (Experimental): The intervention, Tuko Pamoja, is delivered by lay counselors and through existing community social structures, focuses on improving family relationships and mental health with content derived from evidence-based practices; these include solution-focused family therapy and cognitive behavioral strategies. It is components based, with modules delivered based on need. The content and structure has been adapted in both content and implementation model based on formative research in this context. Tuko Pamoja includes a smart phone component to support psychoeducation components and data collection.
  Interventions: Behavioral: Tuko Pamoja, "We are Together" in Kiswahili

INTERVENTIONS:
Behavioral: Tuko Pamoja, "We are Together" in Kiswahili — Tuko Pamoja, "We are Together" in Kiswahili; This intervention, delivered by lay counselors and through existing community social structures, focuses on improving family relationships and mental health with content derived from evidence-based practices; these include solution-focused family therapy and cognitive behavioral strategies. It is components based, with modules delivered based on need. Tuko Pamoja includes a smart phone component to support psychoeducation components and data collection. The content and structure has been adapted in both content and implementation model based on formative research in this context.

SUMMARY:
The purpose of this study is to evaluate a family counseling intervention, entitled "Tuko Pamoja" (Translation "We are Together" in Kiswahili). The intervention, delivered by lay counselors and through existing community social structures, is expected to improve family functioning and individual mental health among members. The sample includes highly distressed families with a child or adolescent (ages 8-17) exhibiting emotional or behavioral concerns; as such, particular emphasis is placed on adolescent-focused outcomes, including mental health and well-being.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a family counseling intervention, entitled "Tuko Pamoja" (Translation "We are Together" in Kiswahili), using a single case series design.

The intervention, delivered by lay counselors and through existing community social structures, focuses on improving family relationships and mental health with content derived from evidence-based practices; these include solution-focused family therapy and cognitive behavioral strategies. It is components based, with modules delivered based on need. The content and structure has been adapted in both content and implementation model based on formative research in this context. Primary hypotheses include achieving improvements in outcomes related to:

1. Family functioning, including elements such as communication, emotional closeness, structure and organization, and satisfaction for the overall family; this also includes indicators of functioning at dyadic levels (i.e., parent-child and couples functioning)
2. Mental health of both children and caregivers, including positive well-being, with a particular emphasis on outcomes for children and adolescents.

The investigators also hypothesize feasibility and acceptability based on a previous evaluation of the program and are analyzing community-sourced practices used by lay counselors. Investigators hypothesize that they are integrating locally-grounded strategies that may influence the delivery or outcomes of the intervention.

The study will follow a single case series design with a sample size of 8 families, including up to 3 caregivers per family (who hold primary responsibility for the child whether biological or non-biological) and a target child identified through caregiver-report of the child about whom they are most concerned. This design will allow for tracking changes in outcome variables over time and for linking clinical changes to session content and delivery strategies.

ELIGIBILITY:
Inclusion Criteria:

* Family with self-reported elevated distress (e.g., high levels of conflict) that also has a child/adolescent (ages 8-17) with caregiver-reported emotional or behavioral concerns

Exclusion Criteria:

* Families without reported distress and/or without reported adolescent distress.
* Families with children older than 17 or younger than 8 years of age.
* Families in which primary caregivers or children are living too far outside of the community to participate in treatment.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Family Functioning: Survey Measure (Change over time) | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  30 self-report items developed for the local context based on formative research. Responses are endorsed on a 10-point scale and refer to the past month. One composite score is calculated; higher scores reflect better family functioning. A subset of these are administered repeatedly pre- and post-intervention as part of the single case series design multiple assessments.
Family Functioning: Direct Observation (Change over time) | Baseline and 1 month post-intervention
  A direct observational measure in which families complete standardized video-recorded activities. Behaviors are then coded on multiple domains, including ones related to positive/negative interactions, quality of communication, and problem-solving ability. Primary analyses will be conducted with higher scores indicating better functioning.
Parent-Child Relationship (Change over time) | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Parent-Child Relationship: from standardized scales and locally developed items. Items selected and adapted from: (1) Parental Acceptance and Rejection Questionnaire, (2) Multiple Indicators Cluster Survey: Discipline Module, (3) Discipline Interview, (4) Parent-Adolescent Communication Scale. Each include caregiver and child/adolescent report versions. Caregiver report includes 66 items; Child report includes 60 items. Participants are asked to respond based on the past month. Children report on each caregiver separately.
  For primary analyses, one composite score will be calculated. For follow-up analyses, subsets of items may be analyzed, including those related specifically to harsh treatment/abuse.
  A subset of these are administered repeatedly pre- and post-intervention as part of the single case series design multiple assessments.
Couples Relationship (Change over time) | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Locally-derived items and selected items adapted from standardized scales: Conflict Tactics Scale; Dyadic Adjustment Scale; additional locally-derived items. A total of 52 items are included, referring to both self and spouse behaviors. The majority of items are based on a frequency scale, referring to the past month; some items related to spousal maltreatment assess whether behaviors have ever occurred.
  As a primary outcome, responses across these items will be combined into one score. Follow-up analyses may be conducted using subsets of items to assess relationship quality and harsh treatment separately.
  A subset of these are administered repeatedly pre- and post-intervention as part of the single case series design multiple assessments.
Child / Adolescent Mental Health (Change over time) | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Items locally developed and adapted from standardized measures, including the Youth Self Report (YSR) and the Child Behavior Checklist (CBCL; for caregivers); locally-developed items assessed local terms reflecting symptoms, hope, prosocial behavior, risk behavior, and sense of belongingness. The majority of items reported on a 3-point scale (Not/Never True, Somewhat/Sometimes True, Very/Often True). Caregiver-report on child included 47 items; Child self-report included 56 items. A single composite score will be calculated, with potential follow-up analyses on subsets of items.
  A subset of these are administered repeatedly pre- and post-intervention as part of the single case series design multiple assessments.
Caregiver Mental Health (Change over time) | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Locally-developed items and items adapted from subscales of standardized measures, including: Patient Health Questionnaire, General Health Questionnaire. Caregivers self-report on 29 total items. One composite score will be calculated, and potential follow-up analyses may examine subsets of items.
  A subset of these are administered repeatedly pre- and post-intervention as part of the single case series design multiple assessments.
Self-defined "Top Problem": Family (Change over time) | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Each participant identifies the two highest priority problems related to their family that they would like the intervention to help with. Items assess how much each problem has bothered them in the past month. For repeated measures as part of the single case series design, these are also administered with participants reporting on the past 2-3 days.
Self-defined "Top Problem": Self (Change over time) | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Each participant identifies the highest priority problem related to themself that they would like the intervention to help with. An item assesses how much the problem has bothered them in the past month. For repeated measures as part of the single case series design, these are also administered with participants reporting on the past 2-3 days.
Self-defined "Top Problem": Child (Change over time) | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Each caregiver identifies the highest priority problem related to their child that they would like the intervention to help with. An item assesses how much the problem has bothered them in the past month. For repeated measures as part of the single case series design, these are also administered with participants reporting on the past 2-3 days.

SECONDARY OUTCOMES:
Counselor Implementation Outcomes | Through study completion
  This measure will assess feasibility, acceptability, and quality of delivery model.
  Fidelity (Checklists, session transcript analysis) Lay counselor competency (session transcript ratings; Adapted ENACT), including counselor use of community practices (session transcript analysis)
  A composite score will be calculated, and follow-up analyses may examine subsets of items dividing fidelity and competency scores.
Material Resources: Household Assets/Consumption (Change over time) | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  This measure includes an inventory of locally-relevant household assets and a measure of consumption and spending. For repeated measures as part of the single case series design, these are also administered with participants reporting on the past 2-3 days.
Alcohol Use: Adult (Change over time) | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  AUDIT (Alcohol Use Disorders Identification Test) and locally-derived items; single items related to associated risk behaviors, such as other substance use, also included. Caregivers self-report on 37 items and spouse-report on 32 items. The majority of items are reported on a frequency Likert scale. Higher scores indicate higher severity.
  For repeated measures as part of the single case series design, these are also administered with participants reporting on the past 2-3 days.
Adolescent Risk Behavior (Change over time) | Baseline and 1 month post-intervention
  Sexually active (Yes/No); Sex past month; Condom use; Number partners; Locally-derived items on peer influence related to risky behaviors
  One risk behavior composite will be calculated, and subsets or single items may be analyzed in follow-up analyses.
Traumatic stress symptoms: Child/Adolescent (Change over time) | Baseline and 1 month post-intervention
  CRIES (Children's Revised Impact of Events Scale), self-reported experience of traumatic stress symptoms over the past week; 8 items (frequency scale). Higher scores indicate higher severity. (These items will be administered if a child endorses 1 or more experiences on the UCLA trauma exposure scale, self-reported experience of traumatic events; 16 items(yes/no)).
Parent-Child Communication: Sex/HIV-Related (Change over time) | Baseline and 1 month post-intervention
  Survey items assessing frequency (6 items) and quality (6 items) of sex/HIV-related communication. Higher scores indicate better communication.
Extended family relationships (Change over time) | Baseline and 1 month post-intervention
  Locally-derived items on quality of relationships with both maternal and paternal extended family members, including positive and negative interactions, as well as any financial or logistical support received. Items are rated on a scale of 1-10. Caregivers report on 10 items; Children report on 6 items. Higher scores indicate better relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Eve S Puffer, PhD, Principal Investigator — Duke University
Locations (1):
- Moi University, Eldoret, Uasin Gishu County, Kenya